CLINICAL TRIAL: NCT00363246
Title: Characterizing Wheelchair-Related Falls in Elderly Veterans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: E4460-R
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Accidental Falls
Keywords: Elderly; Fall risk; Veterans; WheelChairs; Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Older veterans who use a wheelchair for their primary means of mobility.

SUMMARY:
The purpose of this study is to find out about the risk factors for wheelchair-related falls among elderly veterans, and to find out about the costs and consequences of those falls.

DETAILED DESCRIPTION:
Rationale and Objectives. A multitude of risk factors for falls has been reported, however many of these risk factors are not applicable to persons who use a wheelchair for mobility. Specific objectives include: (1) Describe the incidence and prevalence of wheelchair tips (near falls), falls, and fall-related injuries, (2) Describe the epidemiology of the wheelchair tip or fall event. (3) Create models for predicting wheelchair tips, falls, and fall-related injuries for elderly persons who use a wheelchair for mobility. (4) Determine healthcare utilization and direct costs associated with wheelchair-related fall injuries. (5) Describe patient perceived short- and long-term consequences of wheelchair-related falls.

Research Design. This 3-year prospective cohort study includes qualitative and quantitative data collected at baseline data and through monthly follow-up phone interviews over a 12-month period. Data Source. Baseline data on demographics, intrinsic risk factors, and extrinsic risk factors will be collected through interviews. We will assess functional status, cognition, and home management skills through standardized tools. Administrative databases will be used to gather data regarding comorbidities, Veterans Health Administration (VHA) health care utilization and direct costs. A physical therapy assistant will also conduct a wheelchair inventory and wheelchair skills test. Monthly follow-up phone interviews will include number of falls, description of the fall event/mechanism and nature of the injury, changes in modifiable risk factors, and description of injury and treatment. A separate phone interview will be conducted with a subset of subjects at 6 months post fall, using open-ended questions to gather data about patient-perceived long-term consequences of falls. At the end of the 12-month data collection, we will reassess patient's functional status and cognition. Sample. Inclusion criterion includes all veterans who (1) are aged 62 and older, (2) use a wheelchair for their primary means of mobility, (3) have used a wheelchair for at least 12 months previous to enrollment, and (4) will be using a wheelchair for at least the next 12 months. Exclusion criteria (1) no longer living in a community-based setting (e.g., admitted to nursing home), (2) do not have a telephone. We will over sample women and minorities. A total of 882 subjects are needed for a power of 0.8 and an alpha of 0.05 with an anticipated drop out rate of 30%. Analysis. Bivariate analysis will be performed to determine relationships between outcomes and risk factors. Logistic regression models for predicting wheelchair-related tips, falls and fall-related injuries will be developed based on the most important intrinsic and extrinsic risk factors, controlling for possible confounders. Falls will also be analyzed according to a survival-analysis technique. Univariate and multiple Cox regression will be used to assess the associations of different independent variables with the injurious fall. The cost analysis estimates the net or marginal costs of wheelchair users who experience a wheelchair fall accident and seek medical advice or treatment. We use a dichotomous fall (generating medical expense) variable for a "with" or "without" analysis to compare the average cost of medical care for wheelchair users without a fall involving medical observation or care to the average cost of those that did have a serious fall (including death). The difference between these two groups is a proxy of the cost of utilization due to the fall. Multivariate regression analysis will be used to gauge the net effects of a fall on costs, controlling for the wider array of factors that drive cost of treatment and thereby potentially confound univariate analysis. The control variables are demographic including co-morbid conditions and healthcare related.

Anticipated Impact. Our project is expected to identify previously unaccounted for factors that predispose persons who use a wheelchair to falls and fall-related injuries. We will create models for predicting wheelchair tips, falls, and fall-related injuries. These models will be used to develop an evidence-based, patient centered wheelchair falls prevention program targeting modifiable risk factors. Findings from this study will be so used to develop an instrument to identify fall risk in elderly wheelchair users as well as an evidenced-based prevention program. We will partner with the VA National Center for Patient Safety to disseminate these products nationally in the VHA.

ELIGIBILITY:
Inclusion Criteria:

* veteran
* aged 62 and older
* use a wheelchair for their primary means of mobility
* have used a wheelchair for at least 12 months previous to enrollment
* will be using a wheelchair for at least the next 12 months

Exclusion Criteria:

* not living in a community-based setting
* no access to a telephone

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly wheelchair users
Sampling Method: Probability Sample
Enrollment: 766 (Actual)
Dates: Start 2007-06; Primary Completion 2009-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Spehar, DVM MPH JD, Principal Investigator — VA Central Office - HSR&D, Washington, DC
Locations (2):
- James A. Haley Veterans Hospital, Tampa, Florida, United States
- VA Medical Center, San Juan, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 06/01/2007; recruitment ended 11/30/2008. Data collection ended in December 2009. Subjects were approached in a VA medical clinic and given list of qualifying criteria on our flyer. After consent, a Mini-Mental State Examination (MMSE) is administered to all potential subjects; a score of at least 24 is required to participate.
Period: Overall Study
Arm/Group | Group 1
Started | 766
Completed | 669
Not Completed | 97
Not completed — Death | 40
Not completed — Withdrawal by Subject | 19
Not completed — Lost to Follow-up | 14
Not completed — Bad health | 6
Not completed — Stopped using wheelchair | 11
Not completed — Subject expressed security concerns | 2
Not completed — Eligibility changed due to Hospice move | 5

BASELINE CHARACTERISTICS:
Population: Only data for 710 participants for some of the Baseline characteristics.
Arm/Group | Group 1
Number analyzed (Participants) | 766
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 92
  >=65 years | 674
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 738
Race/Ethnicity, Customized [Number; unit: participants] — The data below was subject self-report on baseline survey: "What category best represents your race/ethnicity? (check one) White, Black/African American, Hispanic, etc." Therefore, the racial and ethnic categories must be summed and the totals of racial and ethnic categories will not be equal.
  participants
    Hispanic | 231
    American Indian | 1
    Black or African American | 40
    White | 492
    Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 766
Health [Number; unit: participants] — Participants were asked to characterize their health: Excellent, Very good, good, fair, poor.
  participants
    Excellent/Very Good/Good | 283
    Fair/Poor | 427
    Insufficient data to analyze | 56
Pain in last 4 weeks (interference with daily activities) [Number; unit: participants] — Pain in last 4 weeks and its interference with daily activities
  participants
    None/Mild | 210
    Moderate/Severe | 499
    Missing | 1
    Insufficient data to analyze | 56
Pain when transfer [Number; unit: participants]
  Mild | 315
  Moderate | 180
  Severe | 213
  Missing | 2
  Insufficient data to analyze | 56
Energy levels [Mean (Standard Deviation); unit: units on a scale] — Scale range 4.0-20. Highest energy level = 20.0.
  units on a scale | 11.9 (4.5)

OUTCOME MEASURES:

1. Secondary Outcome: Injuries From Wheelchair-related Falls
Description: Wheelchair-related falls that resulted in an injury in the one year follow up period
Time Frame: one year follow-up period
Population: Older veterans who use a wheelchair for their primary means of mobility. Analyzed for wheelchair-related fall injury during 1-year follow-up period.
Measure: Number; unit: participants
Groups:
- Wheelchair-using Veterans: Older veterans who use a wheelchair for their primary means of mobility. 1 year follow-up period.
Arm/Group | Wheelchair-using Veterans
Number analyzed (Participants) | 710
participants
  No Wheelchair-related fall injuries | 607
  Wheelchair-related fall injuries | 103
Statistical Analysis 1: Comparison: Wheelchair-using Veterans; Health Status. No Wheelchair-related Fall Injuries vs. Wheelchair-related Fall Injuries; Test type: Superiority or Other; p = 0.049, Chi-squared
Statistical Analysis 2: Comparison: Wheelchair-using Veterans; Pain in last 4 weeks (interference with daily activities). No Wheelchair-related Fall Injuries vs. Wheelchair-related Fall Injuries; Test type: Superiority or Other; p = 0.013, Chi-squared
Statistical Analysis 3: Comparison: Wheelchair-using Veterans; Pain when transfer. No Wheelchair-related Fall Injuries vs. Wheelchair-related Fall Injuries; Test type: Superiority or Other; p = 0.0001, Chi-squared
Statistical Analysis 4: Comparison: Wheelchair-using Veterans; Energy level. No Wheelchair-related Fall Injuries vs. Wheelchair-related Fall Injuries; Test type: Superiority or Other; p = 0.009, t-test, 2 sided

2. Primary Outcome: Wheelchair-related Falls
Description: Wheelchair-related falls in 1 year follow-up period.
Time Frame: one year follow-up period
Population: Older veterans who use a wheelchair for their primary means of mobility.
Measure: Number; unit: participants
Arm/Group | Wheelchair-using Veterans
Number analyzed (Participants) | 710
participants
  No Wheelchair-related Fall | 545
  Wheelchair-related Fall | 165
Statistical Analysis 1: Comparison: Wheelchair-using Veterans; Health Status. No Wheelchair-related Falls vs. Wheelchair-related Falls; Test type: Superiority or Other; p = 0.033, Chi-squared; We used chi-squared test for categorical variable (most variables) and t-test (2-sided) for continuous variables (few variables)
Statistical Analysis 2: Comparison: Wheelchair-using Veterans; Pain in last 4 weeks (interference with daily activities). No Wheelchair-related Falls vs. Wheelchair-related Falls; Test type: Superiority or Other; p = 0.013, Chi-squared
Statistical Analysis 3: Comparison: Wheelchair-using Veterans; Pain when transfer. No Wheelchair-related Falls vs. Wheelchair-related Falls; Test type: Superiority or Other; p < 0.001, Chi-squared
Statistical Analysis 4: Comparison: Wheelchair-using Veterans; Energy level. No Wheelchair-related Falls vs. Wheelchair-related Falls; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The original study (PI: Dr. Nelson, Co-PI: Dr. Groer) was approved by the affiliate University of South Florida Institutional Review Board (IRB) on 06/09/2006. Subject recruitment ended November 30, 2008. Data collection ended in December 2009.
Description: This was a non-interventional, observational study of elderly veterans who regularly used a wheelchair for mobility. Adverse events other than death were not collected. Sometimes we were told of a death by a relative when we called. Any serious adverse events were unrelated to the study, which did not involve an intervention.
Groups:
- Elderly Veterans Using Wheelchairs for Mobility: Older veterans who use a wheelchair for their primary means of mobility. This was an observational study. There was no intervention and thus no adverse events were collected as part of the study. Sometimes we learned of a death from a relative when we called monthly.
Arm/Group | Elderly Veterans Using Wheelchairs for Mobility
Serious Adverse Events (participants affected / at risk) | 40/762
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elderly Veterans Using Wheelchairs for Mobility (N=762)
Death (General disorders) | 40 — Subjects were elderly, used a wheelchair, and often had multiple comorbidities, so some deaths during 1-year follow-up could be expected and were unrelated to this observational study. Death note in the computerized medical record or by relative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes